CLINICAL TRIAL: NCT06951022
Title: The Effect of Sujok Therapy on Urinary Incontinence and Quality of Life in Postmenopausal Women
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Gülçin NACAR, Associate Professor, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024/5494
Record Dates: First submitted 2025-04-11; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence (UI); Postmenopause
Keywords: Su Jok Therapy; Urinary Incontinence; Quality of Life; Postmenopausal Women
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants in the experimental group will receive Su Jok seed therapy using apple seeds applied to the hand point that reflects the bladder. Participants will be trained to perform the therapy themselves and will apply it daily for 15 days. They will be reminded via daily messages and monitored for adherence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will receive seed therapy using apple seeds applied to specific hand points corresponding to the bladder area.
  Interventions: Other: Sujok therapy
- Control (No Intervention): standard care

INTERVENTIONS:
Other: Sujok therapy — Participants in the intervention group will receive seed therapy using apple seeds applied to specific hand points corresponding to the bladder area.
  Arms: Intervention

SUMMARY:
This study aims to investigate the effect of Su Jok therapy, a complementary medicine practice, on urinary incontinence and quality of life among postmenopausal women. A total of 120 participants will be included in the study, with 60 in the intervention group and 60 in the control group. Participants in the intervention group will receive Su Jok seed therapy applied to the hand reflex points corresponding to the bladder. The therapy will be administered by the researcher and then taught to the participants, who will continue the application for 15 days. Assessments will be conducted at baseline, day 15, and day 30 using validated questionnaires.

ELIGIBILITY:
Inclusion Criteria:

Women under 65 years of age in the postmenopausal period, Literate, No speech or communication impairment

Exclusion Criteria:

Use of diuretics

Presence of nephrotic syndrome

Diagnosis of diabetes or hypertension

Symptoms of urinary tract infection

Diagnosis of psychiatric illness

History of urinary tract surgery

Diagnosed urinary prolapse

Failure to complete the intervention

Max Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — postmenopausal women
Enrollment: 120 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in urinary incontinence symptoms measured by the International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | At baseline, 15 days and 30 days after intervention
  Description: The ICIQ-SF is a 4-item questionnaire used to evaluate the severity and impact of urinary incontinence.
  Scoring: Scores range from 0 to 21, with higher scores indicating more severe urinary incontinence.
  Unit of Measure: Points on a scale
Change in quality of life measured by the Incontinence Quality of Life Scale (I-QOL) | At baseline, 15 days and 30 days after intervention
  Description: The I-QOL assesses quality of life, including behavioral limitation, psychosocial impact, and social isolation, in postmenopausal women with urinary incontinence.
  Scoring: Domain scores range from 0 to 100, where higher scores represent a poorer quality of life.
  Unit of Measure: Total score (0-100)

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Battalgazi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol